CLINICAL TRIAL: NCT00496067
Title: An Evaluation of a Doppler-Guided Uterine Artery Occlusion Device as Treatment for the Reduction of Fibroid-Associated Bleeding
Brief Title: Uterine Artery Occlusion for Fibroid Related Bleeding
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data required further pilot work to be undertaken.
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Judi Gauld, Manager Clinical Research, Ethicon Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300-06-008
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Menorrhagia; Uterine Fibroids
Keywords: Fibroids; Menorrhagia; Menorrhagia associated with uterine fibroids
MeSH Terms: conditions — Menorrhagia; Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): DUAO Device
  Interventions: Device: Doppler-Guided Uterine Artery Occlusion Device

INTERVENTIONS:
Device: Doppler-Guided Uterine Artery Occlusion Device — For bilateral occlusion of the uterine arteries
  Other Names: floSTAT

SUMMARY:
The primary objective of this study is to evaluate the safety and effectiveness of Doppler guided Uterine Artery Occlusion (D-UAO) as treatment for the reduction of fibroid-associated symptoms.

DETAILED DESCRIPTION:
DUAO is intended for bilateral occlusion of the uterine arteries

ELIGIBILITY:
Inclusion Criteria:

* 25 to 50 years of age
* Subject has a negative urine or blood pregnancy test prior to the procedure. At the time of enrollment to the study, the subject has no intent of further childbearing and intends to use appropriate contraception throughout the first 12 months of the study period (unless sterilized)
* Normal pap smear within 36 months of study procedure (most recent)
* Cervix suitable for tenaculum placement as determined by pelvic exam (adequate length of cervix, absence of cervical fibroid/lower fibroid to prevent clamp placement)
* At least one intra-mural or sub-serosal or sub-mucosal uterine fibroid with a minimum diameter of greater than or equal to 3 cm, and all fibroids with a diameter less than or equal to 8cm with a prevailing pathology (e.g., as opposed to adenomyosis) of fibroids determined through ultrasound
* Symptomatic subject presenting with at least one of the following fibroid symptoms: pelvic pressure, menorrhagia, metrorrhagia, pelvic pain, increasing abdominal girth or dyspareunia due to fibroids.
* Subject has evidence of bilateral ureteric flow
* Subject agrees to participate in the study, including completion of all study-related procedures and evaluations, and documents this agreement by signing the Ethics Committee-approved informed consent.

Exclusion Criteria:

* Pregnancy as confirmed by positive urine or blood pregnancy test
* Menopausal as defined by elevated follicle-stimulating hormone (FSH) and decreased oestradiol hormone levels as determined by the hospital local laboratory reference range criteria
* Presence of any pedunculated sub-mucosal or pedunculated sub-serosal fibroid(s) as determined by MRI, ultrasound or hysteroscopy
* Presence of an intra-uterine device (IUD)
* Any hydronephrosis as determined on renal ultrasound prior to the procedure
* Clinical history of any thrombo-embolic disease or known thrombophilia
* Blood Urine Nitrogen (BUN) greater than 7.2mmol/L* and/or serum creatinine greater than 106μmol/L* unresolved with change in diet or hydration
* History or current evidence of gynecologic malignancy (confirmed by hysteroscopy or endometrial biopsy), atypical endometrial hyperplasia, or chronic pelvic inflammatory disease
* Pelvic mass outside the uterus other than uterine fibroids
* Any current acute or chronic systemic infection or localized pelvic infection, including a urinary tract infection
* Use of Gonadotropin-Releasing Hormone (GnRH) agonist, danozol or mifepristone within 6-months prior to the start of the study procedure
* Using anticoagulation therapy (except over the counter treatments (e.g. aspirin)), or have an underlying bleeding disorder
* Unsuitable for MRI examination (e.g. severe claustrophobia, non-MRI-compatible implanted metalloid devices)
* Prior endometrial ablation, uterine artery embolization, or uterine artery ligation
* Poor procedural candidate due to medical conditions as determined by the investigator (e.g. anesthesia class, renal insufficiency, heart disease);

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2007-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Lack of surgical re-intervention | Post-op through end of study

SECONDARY OUTCOMES:
Percentage of subjects with improvement in Uterine Fibroid Symptom Quality of Life (UFS-QOL) Symptom Severity and Health Related Quality of Life (HRQL) scores. | 6, 12 and 24 months
Mean improvement in UFS-QOL Symptom Severity and HRQL transformed scores. | 6, 12 and 24 months
Mean HRQL subscales. | 6, 12 and 24 months
Percentage of subjects with reduction of 50% or greater in Pictorial Blood Loss Assessment Chart (PBLAC) score. | 6 and 12 months
Mean change in PBLAC scores. | Baseline to 6 and 12 months
Percentage of subjects with decrease in fibroid load based on independent MRI review. | 6 months
Percentage of subjects with maintenance of menses as defined by continuation of menstrual cycles without an interruption of three consecutive months | 12 months
Percentage of subjects with procedural satisfaction as defined by responses of either satisfied or very satisfied. | 12 months
Lack of surgical re-intervention. | 24 months
Pain score | Discharge or 24-hour post clamp removal, whichever is earlier
Days to normal activities (household, work and sexual intercourse) | Post procedure
Euro-QOL expressed as change from baseline for each of the 6 domains and Visual Analogue Scale (VAS) | 1, 3, 6 and 12 months
Nights in hospital | Total and post procedure

CONTACTS AND LOCATIONS:
Overall Officials: David Robinson, MD, Study Director — Ethicon, Inc.
Locations (14):
- Viborg County Hospital, Viborg, Denmark
- France (4):
  - University Hospital, Angers
  - Service de Gynecologie Obsterique, Hopital Antoine Beclere, Clamart
  - Maternite les Bazennes, Dunkirk
  - CHRU de Lille, Hopital Jeanne de Flandre, Lille
- Germany (2):
  - Universitaeklinikum Erlangen, Erlangen
  - Universitats-Frauenklinik Tubingen, Tübingen
- VU Medical Center, Amsterdam, Netherlands
- Ullevaal University, Oslo, Norway
- Universitats-Frauenklinik, Bern, Switzerland
- United Kingdom (4):
  - M1 Maternity, Bradford Royal Infirmary, Bradford
  - Hull and East Yorkshire Women & Children Hospital, Hull
  - Elizabeth Garret Anderson Hospital, London
  - Queen Elizabeth the Queen Mother Hospital, Margate